CLINICAL TRIAL: NCT04138290
Title: A Prospective Post Marketing Surveillance Study Study for the Evaluation of the Safety and Efficacy of the Predictix Antidepressant (PAD) Clinician Software Support Tool in Prescribing Antidepressant Medication/s for the Treatment of Patients Suffering From Major Depressive Disorder
Brief Title: Post Marketing Study for the Evaluation of Predictix Antidepressant Clinician Software Support Tool in Prescribing Antidepressant Medication/s for the Treatment of Patients Suffering From Major Depressive Disorder
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Taliaz Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CL-01-IBR-02
Record Dates: First submitted 2019-10-16; First posted 2019-10-24 (Actual); Last update posted 2019-10-24 (Actual); Status verified 2019-10

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Intervention Model Description: The study is designed as an open label, one arm study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Predictix Antidepressant Software tool (Experimental): Predictix Antidepressant Software tool will be used when prescribed with a medication for their MDD, by their treating physician.
  Interventions: Device: Predictix Antidepressant Software tool

INTERVENTIONS:
Device: Predictix Antidepressant Software tool — Predictix Antidepressant is a stand-alone software tool based on a patients' genetic panel, clinical, demographic and behavioral inputs, intended to support a clinician in choosing the most suitable antidepressant treatment/s for an individual patient diagnosed with Major Depressive Disorder.

SUMMARY:
The study is designed as an open label, one arm study. Up to 30 eligible patients will be enrolled, for whom the Predictix Antidepressant Software tool will be used when prescribed with a medication for their Major Depressive Disorder, by their treating physician.

Visits will include the completion of several questionnaires designed to answer the study objectives, either as self-reported by the subjects and/ or by the clinician.

DETAILED DESCRIPTION:
The study will enroll up to 30 eligible patients, for whom the Predictix Antidepressant Software tool will be used when prescribed with a medication for their Major Depressive Disorder, by their treating physician.

A treatment cycle will include four to five visits: Information consent and oral sampling, Baseline, 4 and 8 weeks. At least one completed cycle per patient is required for a patient to be included in the analysis as study completed.

The treating physician will review and approve each subject's eligibility prior to his/ her entrance to the study and will review the Predictix Antidepressant software tool report prior to treatment start.

Visits will include the completion of the Taliaz Ltd. Physician Form and several questionnaires designed to answer the study objectives Usability and satisfaction questionnaire/s will be analyzed for Usefulness, Satisfaction, Ease of Use and Learnability of the system.

ELIGIBILITY:
Inclusion Criteria:

* Male and female at the age of 18 - 75 years old
* Indication of MDD diagnosis per DSM V
* Rule out other causes of depressive symptoms other than MDD apart from General Anxiety Disorder as authentified by the MINI*) (by Sheehan and Lecrubier ).

  *Up to a maximum of 15 completed GAD pts
* Ability to read, understand and sign an informed consent document

Exclusion Criteria:

* Patient is diagnosed with other major psychopathologies (i.e. schizophrenia, bipolar disorder, psychotic depression, geriatric depression)
* Patient requires antipsychotic medication or mood stabilizers
* Patient is at substantial suicidal risk as judged by the treating physician
* Patient has attempted suicide in the past year.
* Patient has any current unstable medical condition or surgical illness
* Patient has history of seizure or convulsions.
* Patient has history of drug abuse or alcoholism in the last 6 months
* Inadequate communication with the patient
* In the investigator's judgement, patient is not able to provide written informed consent
* Pregnant women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-12 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
success rate of the Predictix tool | 8 weeks
  A success will be defined as a score of 3 and below in the total improvement: measured by the CGI last measured value compared to Baseline, as well as a >50% improvement measured by the QIDS16, under a specific medication cycle regimen.

SECONDARY OUTCOMES:
Usability | 8 weeks
  Usability n questionnaire will be analyzed

OTHER OUTCOMES:
To evaluate the effect of device use on patients' care outcomes in terms of economic burden and social impact | 8 weeks
  by analyzing the completed Work Productivity and Activity Impairment (WPAI) questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Pitié Salpétrière, Paris, France

IPD SHARING:
Plan to Share IPD: No